CLINICAL TRIAL: NCT07244978
Title: A Prospective, Single-arm, Single-center, Exploratory Study of the Safety and Efficacy of Ivonescimab（AK112） Combined With Chemotherapy in Patients With Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Ivonescimab（AK112） Combined With Chemotherapy in Patients With Resectable Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1704
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapy
Keywords: ivonescimab; anti-PD-1; anti-VEGF; Neoadjuvant; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy; Esophagectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivonescimab（AK112） Combined With Chemotherapy (Experimental): Preoperative neoadjuvant therapy for 3 cycles. Radical surgery is performed 4-8 weeks after the last dose. Postoperative radiotherapy is determined according to the clinical situation and pathological stage of the patient.
  Ivonescimab（AK112） can be maintained for a maximum of 1 year. During the study, patients were be followed until disease progression, withdrawal of informed consent, loss of follow-up, or death.
  Interventions: Combination Product: Ivonescimab（AK112), Albumin paclitaxel, carboplatin AUC=5, neoadjuvant therapy; Procedure: Esophagectomy; Other: Sample

INTERVENTIONS:
Combination Product: Ivonescimab（AK112), Albumin paclitaxel, carboplatin AUC=5, neoadjuvant therapy — Ivonescimab（AK112) 20mg/kg, IV, Day 1; Albumin paclitaxel 260mg/m2, Day 1; carboplatin AUC=5, Day 1; Preoperative neoadjuvant therapy for 3 cycles, one cycle every 21 days.
Procedure: Esophagectomy — Prior to each surgical procedure, the department engaged in comprehensive discussions and deliberations to ascertain and establish the most suitable course of action. Minimally invasive Ivor-Lewis (intrathoracic anastomosis) or McKeown (neck anastomosis) esophagectomy, including two field extensive lymphadenectomies, was performed according to the tumor location. The resection length should be at least 5cm from the tumor origin according to prechemotherapy by endoscopy.
  The surgeries will be performed by surgeons with rich experience. Minimally invasive esophagectomy, can be performed using the da Vinci surgical robot, thoracoscope, or laparoscope, or by using an open approach, as judged appropriate by the surgeon.
Other: Sample — Blood, Tumour will be Collected from participant. Fate of sample is Destruction after use.
  5 ml of peripheral blood was collected the day before each of the immunotherapy sessions and after surgery.
  Tumour sample will be collected before neoadjuvant therapy and during surgery.

SUMMARY:
In the past few decades, surgery, radiotherapy, chemotherapy and other treatments were continuously improved, however, the mortality of esophageal squamous cell carcinoma patients was not significantly decreased. It is recommended that a treatment strategy be employed that integrates surgery with radiotherapy, chemotherapy, or immunotherapy, in order to enhance overall survival by improving local-regional tumor control and addressing microscopic metastases. Clinical research indicates that combining anti-PD-1/L1 and anti-VEGF antibodies enhances anti-tumor effects in esophageal squamous cell carcinoma. Ivonescimab, a humanized bispecific monoclonal antibody targeting PD-1/VEGF. This single-arm, prospective, exploratory study is planned to evaluate the combination of ivonescimab and chemotherapy in neoadjuvant therapy for resectable esophageal squamous cell carcinoma, with the aim of providing new therapeutic options for this condition.

DETAILED DESCRIPTION:
China with high incidence of esophageal cancer, the number of new cases and deaths account for about 50% of the world every year. In the past few decades, surgery, radiotherapy, chemotherapy and other treatments were continuously improved, however, the mortality of esophageal squamous cell carcinoma patients was not significantly decreased. For patients with locally advanced esophageal squamous cell carcinoma, direct surgery is not effective. It is difficult to achieve radical resection by surgery merely, and even if many patients receive surgery, they may eventually have tumor recurrence and poor survival rate.

It is recommended that a treatment strategy be employed that integrates surgery with radiotherapy, chemotherapy, or immunotherapy, in order to enhance overall survival by improving local-regional tumor control and addressing microscopic metastases. Consequently, the exploration of effective perioperative adjuvant or neoadjuvant treatment modalities aimed at reducing the risk of postoperative recurrence and enhancing postoperative survival rates is a critical focus in the treatment of esophageal squamous cell carcinoma.

Recently, PD-1/ PD-L1 immunocheckpoint inhibitor may become a new method for the treatment of esophageal cancer. Clinical research indicates that combining anti-PD-1/L1 and anti-VEGF antibodies enhances anti-tumor effects in esophageal squamous cell carcinoma. Ivonescimab, a humanized bispecific monoclonal antibody targeting PD-1/VEGF, boosts the immune system's anti-tumor response and inhibits VEGF's immunosuppressive effects, enhancing T cell infiltration in tumors. In patients with locally advanced esophageal cancer, the efficacy of ivonescimab combined with chemotherapy for sequential radical surgery is still unclear. Therefore, a single-arm, prospective, exploratory study is planned to evaluate the combination of ivonescimab and chemotherapy in neoadjuvant therapy for resectable esophageal squamous cell carcinoma, with the aim of providing new therapeutic options for this condition.

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent;
2. patients age 18 to 75 years old
3. primary resectable, histologically confirmed esophageal squamous cell cancer;
4. Esophageal squamous cell carcinoma the clinical stage was II-IVA (according to AJCC TNM stage, 8th edition).
5. ECOG PS 0-1.
6. No distant metastasis, the diseases could be resectable assessed by thoracic oncologist;

Exclusion Criteria:

1. with significant cardiovascular disease;
2. current treatment with anti-viral therapy or HBV;
3. Female patients who are pregnant or lactating;
4. history of malignancy within 5 years prior to screening;
5. active or history of autoimmune disease or immune deficiency;
6. signs of distant metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete response (PCR) | 1 month after surgery
  The proportion of the surgical population with PCR, which was defined no residual invasive tumor cells were found in the pathological examination of resected specimens, including the primary tumor and lymph nodes.

SECONDARY OUTCOMES:
Rate of major pathological response (MPR) | 1 month after surgery
  The proportion of the surgical population with MPR, which was defined in the pathological examination of resected specimens, the proportion of residual tumor cells was less than 10%.
Rate of objective response rate (ORR) | before surgery
  The proportion of subjects with imaging PR or CR assessed according to RECIST 1.1 criteria
2-year and 5-year overall survival rate | 2-year and 5-year after enrolled
  The proportion of all study cases in which no death from any cause occurred within 2 years and 5 years after surgery
Incidence of Treatment-related Adverse Events | 1 month after surgery
  Incidence of Treatment-related Adverse Events as Assessed by CTCAE v5.0
The changes in the peripheral blood immunoprofile and tumor tissue sample among non-PCR (NPCR) and PCR patients | 3 month after surgery
  By using mass spectrometry (CyTOF), single-cell analysis, and other detecting techniques , we comprehensively characterized the immune landscape in the peripheral blood and tumor sample of ESCC patients before and after anti-PD-1 immunotherapy, aiming to explore the immune subsets correlated with neoadjuvant immunotherapy response.

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China